CLINICAL TRIAL: NCT03229135
Title: A Retrospective Study of Relationships Between Loading Regimen，Serum Trough Concentrations，Efficacy and Safety in Pneumonia Patients With Gram-positive Infections Treated With Teicoplanin
Brief Title: Loading Regimen，Serum Trough Concentrations，Efficacy and Safety in Pneumonia Patients With Gram-positive Infections
Status: Completed | Type: Observational
Sponsor: People's Hospital of Zhengzhou University (Other)
Responsible Party: Principal Investigator, LIjuan Zhou, Principal Investigator, People's Hospital of Zhengzhou University
Other Study IDs: LZhou
Record Dates: First submitted 2017-07-19; First posted 2017-07-25 (Actual); Last update posted 2017-07-25 (Actual); Status verified 2017-07

CONDITIONS: Pneumonia Gram-Positive Bacterial

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (4):
- Group A: Group A (CLcr≥60mL/min) : Teicoplanin was intravenously administered 3 times for moderate infections (skin, soft tissue and respiratory infections) or 6 times for severe infections(endocarditis caused by MRSA or severe pneumonia) at the loading dose of 400 mg at 12h intervals, followed by maintenance dosing 400 mg/d.
  Interventions: Device: other antibacterial agents，breathing machine
- Group B: Group B (40 mL/min≤CLcr<60mL/min) : Teicoplanin was intravenously administered 3 times at the loading dose of 400 mg at 12h intervals, followed by maintenance dosing 400 mg/d.
  Interventions: Device: other antibacterial agents，breathing machine
- Group C: Group C (CLcr<40mL/min) : Teicoplanin was intravenously administered 2 times at the loading dose of 400 mg at 12h intervals, followed by maintenance dosing 200 mg/d.
  Interventions: Device: other antibacterial agents，breathing machine
- Group D: Group D (standard regimen) : Teicoplanin was intravenously administered 1-3 times at the loading dose of 400 mg at 12h intervals, followed by maintenance dosing 200 mg/d.
  Interventions: Device: other antibacterial agents，breathing machine

INTERVENTIONS:
Device: other antibacterial agents，breathing machine — If treatment failure for patients in group A，group B，group C and group D，change dose of teicoplanin or other antibacterial agents. Mechanical ventilation was adopte.Treatment failure was defined as no improvement or worse of clinical symptoms, laboratory data, requiring change of teicoplanin therapy.

SUMMARY:
This was a retrospective study that all teicoplanin-treated adult patients with Gram-positive infections admitted to Zhengzhou Central Hospital affiliated to Zhengzhou University from February 2015 to August 2016.

DETAILED DESCRIPTION:
1. Patients and protocol This was a retrospective study that all teicoplanin-treated adult patients with Gram-positive infections admitted to Zhengzhou Central Hospital affiliated to Zhengzhou University from February 2015 to August 2016. Patients were included who met the following criteria: (1) age≥18 years, (2) duration of teicoplanin therapy≥5 days, (3) written informed consent was obtained from each patients. Patients were excluded who fulfilled any of the following criteria: (1) Patients who were allergy to teicoplanin, (2) pregnant women, (3) patients with hematopoietic function, (4) patients unable to evaluate efficacy and safety. This study was approved by the research ethics committee of the Zhengzhou Central Hospital affiliated to Zhengzhou University.
2. Treatment regimen and groups According to CLcr and teicoplanin loading dose regimen, all patients were divided into four groups. Group A (CLcr≥60mL/min) : Teicoplanin was intravenously administered 3 times for moderate infections (skin, soft tissue and respiratory infections) or 6 times for severe infections(endocarditis caused by MRSA or severe pneumonia) at the loading dose of 400 mg at 12h intervals, followed by maintenance dosing 400 mg/d. Group B (40 mL/min≤CLcr<60mL/min) : Teicoplanin was intravenously administered 3 times at the loading dose of 400 mg at 12h intervals, followed by maintenance dosing 400 mg/d. Group C (CLcr<40mL/min) : Teicoplanin was intravenously administered 2 times at the loading dose of 400 mg at 12h intervals, followed by maintenance dosing 200 mg/d. Group D (standard regimen) : Teicoplanin was intravenously administered 1-3 times at the loading dose of 400 mg at 12h intervals, followed by maintenance dosing 200 mg/d. The maintenance dosing was adjusted by Cmin and CLcr in all groups. The target Cmin was set to 15~30 mg/L. If Cmin<15 mg/L or >30 mg/L, the maintenance dosage was increased or decreased appropriately up to target Cmin range. CLcr values for male and female were calculated based on the following equations, respectively.

ELIGIBILITY:
Inclusion Criteria:

* age≥18 years
* duration of teicoplanin therapy≥5 days
* written informed consent was obtained from each patients

Exclusion Criteria:

* Patients who were allergy to teicoplanin
* pregnant women
* patients with hematopoietic function
* patients unable to evaluate efficacy and safety

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The clinical data of 113 patients who were suffered with severe Gram-positive infection and treated with teicoplanin from February 2015 to August 2016 were retrospectively analyzed.
Sampling Method: Non-Probability Sample
Enrollment: 113 (Actual)
Dates: Start 2015-02-01 (Actual); Primary Completion 2016-08-20 (Actual); Study Completion 2016-10-30 (Actual)

PRIMARY OUTCOMES:
Serum teicoplanin trough concentrations | 0.5 hour before teicoplanin administration on the fourth day
  Teicoplanin trough samples were taken immediately 30 minutes before teicoplanin administration on the fourth day. Blood samples for 2-3 mL were collected in blood-collection tubes without any additives and centrifuged at 3500 rpm for 10min. Serum teicoplanin trough concentrations (Cmin) were determined by a high-performance liquid chromatography method as previously described. The detections were completed in Translational Medicine Center of Zhengzhou Central Hospital affiliated to Zhengzhou University.

SECONDARY OUTCOMES:
White blood cell count (WBC) | 2 years
  It was completed before initiation and after completion of teicoplanin therapy in Zhengzhou city clinical inspection center.
C-reaction protein (CRP) | 2 years
  It was completed before initiation and after completion of teicoplanin therapy in Zhengzhou city clinical inspection center.
Asparttate aminotransferase (AST) | 2 years
  It is an indicator of liver function.It was completed before initiation and after completion of teicoplanin therapy in Zhengzhou city clinical inspection center.
Alanine aminotransferase (ALT) | 2 years
  It is an indicator of liver function.It was completed before initiation and after completion of teicoplanin therapy in Zhengzhou city clinical inspection center.
Serum creatinine (Scr) | 2 years
  It is an indicator of renal function.It was completed before initiation and after completion of teicoplanin therapy in Zhengzhou city clinical inspection center.
CLcr | 2 years
  It is an indicator of renal function.It was completed before initiation and after completion of teicoplanin therapy in Zhengzhou city clinical inspection center.

IPD SHARING:
Plan to Share IPD: No